CLINICAL TRIAL: NCT06407635
Title: Psilocybin for PTSD With or Without Psychotherapy: A Pilot Study of Safety and Efficacy
Brief Title: A Study of Psilocybin for PTSD
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Steven & Alexandra Cohen Foundation (Other); Usona Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00407008
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trauma-focused psychotherapy treatment condition (Experimental): Individuals in this arm will undergo procedures related to trauma-focused psychotherapy (combined with standard psychological support) beginning after receipt of psilocybin.
  Interventions: Drug: Psilocybin; Other: Trauma-focused psychotherapy; Other: Standard psychological support
- Standard psychological support treatment condition (Active Comparator): This condition represents typical support following the experimental administration of psilocybin therapy.
  Interventions: Drug: Psilocybin; Other: Standard psychological support

INTERVENTIONS:
Drug: Psilocybin — The two psilocybin doses will be administered approximately 2 weeks apart in the form of an oral capsule. The first dose will be 25mg. For the second dosing session, participants will either remain on 25 mg of psilocybin, or will receive a dose of 40 mg, depending on the strength of subjective effects experienced during the first dosing session, as well as clinical judgment and participant preference.
Other: Trauma-focused psychotherapy — Components of trauma-focused psychotherapy will include Cognitive Processing Therapy and in vivo exposure. Such components of evidence-based psychotherapy may lower the safety risk profile for this vulnerable population and enhance the effect size and maintenance of psilocybin therapy.
  Arms: Trauma-focused psychotherapy treatment condition
Other: Standard psychological support — Standard psychological support involves providing a safe and emotionally supportive environment to participants throughout the course of their participation, and being attentive and responsive to their emotional needs. It includes continued review and discussion of experiences that participants encountered during the psilocybin sessions and the way that those experience relate to the participant's life and clinical status.

SUMMARY:
The proposed open-label, controlled study at the Johns Hopkins Center for Psychedelic and Consciousness Research (CPCR) will test the following primary hypotheses in adult patients with chronic PTSD who are currently taking a serotonin reuptake inhibitor: psilocybin therapy will be feasible and safe for participants, significantly remediate PTSD symptoms, and enhance wellbeing and quality of life. In addition, the study will examine whether elements of evidence-based trauma-focused psychotherapy enhance treatment response when paired with psilocybin.

DETAILED DESCRIPTION:
This study uses a randomized controlled design to compare the safety and efficacy of 2 doses of psilocybin for PTSD. In addition, it will investigate the effects of trauma-focused psychotherapy (which includes standard psychological support) versus standard psychological support alone. Twenty participants will be recruited. Following the first psilocybin session, participants will be randomized to either the trauma-focused psychotherapy (which includes standard psychological support) treatment condition or the standard psychological support treatment condition (the latter being typical for the experimental administration of psilocybin therapy). Both groups will receive identical treatment prior to receiving the first dose of psilocybin, with one group receiving procedures related to trauma-focused psychotherapy (combined with standard psychological support) beginning after receipt of psilocybin. The study will include clinician and participant ratings of PTSD and mood symptoms pre- and post-drug session and monitor and participant ratings of subjective drug effects during and after each drug session.

The intervention for both groups will consist of about 8 hours of preparatory meetings (over approximately 2 weeks), followed by 2 psilocybin sessions separated by approximately 2 weeks. The initial psilocybin dose will be 25 mg. The dose for the second session may be increased conditional on the strength of subjective effects, as measured by the Mystical Experiences Questionnaire (MEQ30), taken at the end of participants' first psilocybin session. This allows a dose to increase if, for example, concomitant serotonin reuptake inhibitors reduce subjective effects. Participants with a score ≥60% of the maximum on the MEQ30 will remain at a dose of 25 mg of psilocybin for the second session. Participants with an MEQ30 score below 60% will receive a dose of 40 mg for the second session. Elevation of dose will also be based on the clinical judgment of the principal investigator, study physician, and study staff that a higher dose can be safely administered. In addition, participants who prefer to not elevate the dose will remain at 25 mg for the second session.

To support the participant's therapeutic integration of psilocybin experiences, following each psilocybin session, participants will meet with the session facilitator(s) at multiple scheduled time points. Additional contact hours will be scheduled if it is judged that the participant would benefit from additional meetings to discuss experiences from the session(s) or to prepare for the next session.

This study is supported in part by philanthropic contributions from private individuals. These donors are not involved in the design, conduct, or analysis of the research.

ELIGIBILITY:
Inclusion criteria:

* Be at least 21 years old
* Have given written informed consent
* Have a confirmed DSM-5 diagnosis of Post-Traumatic Stress Disorder with symptom duration >= 6 months
* Have a baseline CAPS-5 score of >=35
* Currently taking a serotonin reuptake inhibitor (SSRI or SNRI) at a stable dose for at least 3 months.
* Be judged by study team clinicians to be at low acute risk for suicidality
* Be medically stable as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests
* Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the mornings of drug session days. If the participant does not routinely consume caffeinated beverages, he/she must agree not to do so on session days.
* Agree to refrain from using alcohol, anxiolytics, stimulants, sedatives or hypnotics, opioids, dissociatives, cannabinoids, or other unapproved substances within 24 hours of psilocybin administration. Caffeine and nicotine are exceptions.
* Agree not to take any as needed (PRN) medications on the mornings of drug sessions
* Agree to stop taking 5HT2A antagonist medications at least 5 half-lives before psilocybin dosing.
* Agree not to take sildenafil (Viagra®), tadalafil, or similar medications within 72 hours of each drug administration.
* Have no classic psychedelic use in the past five years.
* Have at least a high school level of education or equivalent (e.g. GED).
* Weigh at least 40kg.
* (for female participants) Agree to use highly effective birth control measure within two weeks before and after dosing sessions.
* (for male participants) Agree to use contraception and refrain from sperm donation two weeks before and after dosing sessions, as the reproductive safety for psilocybin is not yet established.

Exclusion Criteria:

General medical exclusion criteria:

* Women who are pregnant (as indicated by a positive urine pregnancy test assessed at intake and before each drug session) or nursing; women who are of child- bearing potential and sexually active who are not practicing an effective means of birth control.
* Cardiovascular conditions: coronary artery disease, stroke, angina, hypertension with resting blood pressure systolic >139 or diastolic >89, a clinically significant ECG abnormality (e.g., atrial fibrillation), prolonged corrected QT interval (QTc) interval (i.e., QTc > 450 msec), artificial heart valve, or transient ischemic attack (TIA) in the past year
* Family history of Torsades de Pointes and sudden cardiac death
* Epilepsy with history of seizures
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* Currently taking a Monoamine Oxidase Inhibitor

Psychiatric Exclusion Criteria:

* Current or past history of meeting DSM-5 criteria for schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition), or Bipolar I or II Disorder
* Current or history within one year of meeting DSM-5 criteria for a severe alcohol, tobacco, or other drug use disorder (excluding caffeine)
* Current or history within one year of meeting DSM-5 criteria for Borderline Personality Disorder.
* Have a first degree relative with schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition), or Bipolar I.
* Has a psychiatric condition judged to be incompatible with establishment of rapport or safe exposure to psilocybin
* History of a medically significant suicide attempt
* Unwilling or unable to pause concurrent psychotherapy during the study.
* Determined to be at risk for re-exposure to the index trauma or other significant trauma in daily life.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 8 months
  Adverse event monitoring throughout the study.
Columbia Suicide Severity Rating Scale (C-SSRS) | 8 months
  Used to assess severity of suicide ideation during every study visit. The C-SSRS has a score range of 0-5, with 0 being the least severe and 5 being the most severe. The scale has ten categories, all of which are binary responses (yes/no) that indicate the presence or absence of a behavior.
Clinician-Administered PTSD Scale for Diagnostic and Statistical Manual (DSM)-5 (CAPS-5) | 8 months
  The CAPS-5 assessment consists of 30 items that are designed to measure the frequency and intensity of PTSD symptoms, covering all 20 DSM-5 PTSD symptoms. Each item is scored on a 5-point scale (0-4), with 0 being absent and 4 being extreme/incapacitating. Higher scores indicate higher severity of PTSD symptoms.
Ecological Momentary Assessment (EMA) of PTSD Checklist for DSM-5 (PCL-5) | 3 months
  The PTSD Checklist for DSM-5 (PCL-5; is a self-report psychometric instrument widely employed in both clinical and research settings to assess the presence and severity of PTSD symptoms as outlined in the DSM-5. The PCL-5's 20 items correspond to the DSM-5 symptom criteria for PTSD. For this study, PCL-5 symptoms are assessed using Ecological Momentary Assessment (EMA), such that respondents will be asked to rate the degree to which they have been bothered by each symptom within a preceding time-frame (e.g., preceding 2 hours, preceding day) on a Likert scale ranging from 0 (Not at all) to 4 (Extremely). A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items with higher scores indicating greater symptom severity.
World Health Organization Quality of Life Brief Version (WHOQOL-BREF) | 8 months
  An internationally recognized and validated tool for evaluating an individual's perception of their position in life, within the context of their culture and value system, and relative to their personal goals, expectations, standards, and concerns. Consists of multiple domains and facets, covering physical health, psychological health, social relationships, and environment. Each of these domains is assessed through several questions that the respondent answers on a five-point Likert scale. These scores are then used to compute an overall score, which is transformed linearly to a 0-100-scale with higher scores indicating a better perceived quality of life.

SECONDARY OUTCOMES:
Beck Depression Inventory II (BDI-II) | 8 months
  Used to assess depressive symptoms. BDI-II is scored by adding up the highest ratings for each of the 21 items on the questionnaire, which range from 0 to 3. The total score can range from 0 to 63, with higher scores indicating more severe depressive symptoms.
Sheehan Disability Scale (SDS) | 8 months
  Used to assess functional impairment in three domains of disability that can be impaired during depression: work/school, social, and family life. Total score 0-30 (0 unimpaired, 30 highly impaired) Work/school (0-10) Social life (0-10) Family life/home responsibilities (0-10) Scores of ≥5 on any of the 3 scales; high scores are associated with significant functional impairment.
Posttraumatic Maladaptive Beliefs Scale (PMBS) | 3 months
  This 15-item scale assesses maladaptive beliefs related to PTSD, indexed by three subscales including (1) Threat of Harm, (2) Self-Worth and Judgment, and (3) Reliability and Trustworthiness of Others. Scores on each subscale can be derived by summing items within each subscale. A list of subscale items and reverse-code directions are indicated on the measure. Possible scores range from 15-105, and subscale scores range from 5-35. Higher scores are indicative of more maladaptive beliefs in each of the three domains assessed within this measure.

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Nayak, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Center for Psychedelic and Consciousness Research, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No